CLINICAL TRIAL: NCT06594445
Title: HM2023-05: GTB-3650 (Anti-CD16/IL-15/Anti-CD33) Tri-Specific Killer Engager (TriKE®) for the Treatment of High Risk Myelodysplastic Syndromes (MDS) and Refractory/Relapsed Acute Myeloid Leukemia (AML)
Brief Title: HM2023-05: GTB-3650 Trike for High Risk MDS and R/R AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023LS024
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Myeloid Malignancy; Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm 1: Dose Level 1: 1.25 ug/kg/day (Experimental): GTB-3650 is administered during an inpatient stay by continuous infusion (CI) consisting of three consecutive 24 hour infusion "bags" over a 72 hour period. Each 72-hour infusion period is designated a "block".
  A 28-day treatment cycle consists of two blocks followed by approximately 18 days of no treatment. Prior to each block start, the patient must meet the safety criteria.GTB-3650 may continue for up to four treatment cycles total provided disease based response criteria is met and the patient is otherwise eligible to continue.
  Interventions: Drug: GTB-360
- Arm 2: Dose Level 2: 2.5 ug/kg/day (Experimental): GTB-3650 is administered during an inpatient stay by continuous infusion (CI) consisting of three consecutive 24 hour infusion "bags" over a 72 hour period. Each 72-hour infusion period is designated a "block".
  A 28-day treatment cycle consists of two blocks followed by approximately 18 days of no treatment. Prior to each block start, the patient must meet the safety criteria.GTB-3650 may continue for up to four treatment cycles total provided disease based response criteria is met and the patient is otherwise eligible to continue.
  Interventions: Drug: GTB-360
- Arm 3: Dose Level 3: 5 ug/kg/day (Experimental): GTB-3650 is administered during an inpatient stay by continuous infusion (CI) consisting of three consecutive 24 hour infusion "bags" over a 72 hour period. Each 72-hour infusion period is designated a "block".
  A 28-day treatment cycle consists of two blocks followed by approximately 18 days of no treatment. Prior to each block start, the patient must meet the safety criteria.GTB-3650 may continue for up to four treatment cycles total provided disease based response criteria is met and the patient is otherwise eligible to continue.
  Interventions: Drug: GTB-360
- Arm 4: Dose Level 4: 10 ug/kg/day (Experimental): GTB-3650 is administered during an inpatient stay by continuous infusion (CI) consisting of three consecutive 24 hour infusion "bags" over a 72 hour period. Each 72-hour infusion period is designated a "block".
  A 28-day treatment cycle consists of two blocks followed by approximately 18 days of no treatment. Prior to each block start, the patient must meet the safety criteria.GTB-3650 may continue for up to four treatment cycles total provided disease based response criteria is met and the patient is otherwise eligible to continue.
  Interventions: Drug: GTB-360
- Arm 5: Dose Level 5: 25 ug/kg/day (Experimental): GTB-3650 is administered during an inpatient stay by continuous infusion (CI) consisting of three consecutive 24 hour infusion "bags" over a 72 hour period. Each 72-hour infusion period is designated a "block".
  A 28-day treatment cycle consists of two blocks followed by approximately 18 days of no treatment. Prior to each block start, the patient must meet the safety criteria.GTB-3650 may continue for up to four treatment cycles total provided disease based response criteria is met and the patient is otherwise eligible to continue.
  Interventions: Drug: GTB-360
- Arm 6: Dose Level 6: 50 ug/kg/day (Experimental): GTB-3650 is administered during an inpatient stay by continuous infusion (CI) consisting of three consecutive 24 hour infusion "bags" over a 72 hour period. Each 72-hour infusion period is designated a "block".
  A 28-day treatment cycle consists of two blocks followed by approximately 18 days of no treatment. Prior to each block start, the patient must meet the safety criteria.GTB-3650 may continue for up to four treatment cycles total provided disease based response criteria is met and the patient is otherwise eligible to continue.
  Interventions: Drug: GTB-360
- Arm 7: Dose Level 7: 100 ug/kg/day (Experimental): GTB-3650 is administered during an inpatient stay by continuous infusion (CI) consisting of three consecutive 24 hour infusion "bags" over a 72 hour period. Each 72-hour infusion period is designated a "block".
  A 28-day treatment cycle consists of two blocks followed by approximately 18 days of no treatment. Prior to each block start, the patient must meet the safety criteria.GTB-3650 may continue for up to four treatment cycles total provided disease based response criteria is met and the patient is otherwise eligible to continue.
  Interventions: Drug: GTB-360

INTERVENTIONS:
Drug: GTB-360 — GTB-3650 is administered by a continuous infusion (CI). A patient's dose of GTB-3650 is calculated using their assigned Dose Level and their actual body weight (ABW) obtained within 5 days prior to or on Cycle 1, Day 1.
  Dose Level 1: 1.25 ug/kg/day Dose Level 2: 2.5 ug/kg/day Dose Level 3: 5 ug/kg/day Dose Level 4: 10 ug/kg/day Dose Level 5: 25 ug/kg/day Dose Level 6: 50 ug/kg/day Dose Level 7: 100 ug/kg/day
  Other Names: anti-CD16/IL-15/anti-CD33

SUMMARY:
This is a Phase I dose finding study of GTB-3650 (anti-CD16/IL-15/anti-CD33) Tri-Specific Killer Engager (TriKE®) for the treatment of select CD33-expressing refractory/relapsed myeloid malignancies in adults ≥ 18 years of age who are not a candidate for potentially curative therapy, including hematopoietic stem cell transplantation, and are refractory to, intolerant of, or ineligible for therapy options that are known to provide clinical benefit. The hypothesis is GTB-3650 TriKE will induce natural killer (NK) cell function by targeting malignant cells, as well as, CD33+ myeloid derived suppressor cells (MDSC) which contribute to a tumor induced immunosuppression. Because CD16 is the most potent activating receptor on NK cells, this single agent may induce a targeted antiCD33+ tumor response

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a high risk myelodysplastic syndromes (MDS), treatment related MDS, OR relapsed/refractory acute myelogenous leukemia (AML).
* Absolute lymphocyte count (ALC) ≥ 200 cells/µL OR absolute circulating CD56+/CD3- NK cell count >25 cells/µL within the 14 days prior to Cycle 1 Day 1.
* Peripheral blasts ≤20,000 at the time of treatment start. Hydroxyurea may be used up to Day 1 of the 1st cycle to achieve this threshold and continued for the 1st two weeks of Cycle 1 to maintain it.
* Karnofsky performance status ≥ 70%
* Adequate organ function within 14 days (30 days for cardiac) of Cycle 1 Day 1
* Sexually active persons of childbearing potential or persons with partners of childbearing potential must agree to use a highly effective form of contraception during study treatment and for at least 4 months after the last dose of GTB-3650. Non-childbearing is defined as >1 year postmenopausal or surgically sterilized.

-For the Dose Finding Component Only: Must agree to stay within a 60- minute drive of the Study Center through the Cycle 1 Day 29 visit (end of the Dose Limiting Toxicity period).

* Provides voluntary written consent prior to the performance of any research related activity.
* Pulmonary: room air 0 2 saturation at ≥ 95%

Exclusion Criteria:

* Pregnant or breast-feeding. The effect of GTB-3650 TriKE on the fetus is unknown. Persons of childbearing potential must have a negative serum or urine test within 7 days prior to Cycle 1 Day 1 to rule out pregnancy.
* A candidate for hematopoietic stem cell transplant (HSCT) or newly relapsed after HSCT (e.g. no post-HSCT therapy given).
* Bi-phenotypic acute leukemia or mixed lineage leukemia.
* Acute promyelocytic leukemia (APL).
* No anticancer therapy within 14 days of Cycle 1 Day 1; any AEs from therapy given prior must have resolved to Grade 1 or baseline
* New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving with associated clinical improvement after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Active systemic infection requiring parenteral antibiotic therapy. Any prior systemic infections must have resolved following optimal therapy.
* Known history of HIV.
* Active Hepatitis B or Hepatitis C (virus detectable by PCR) - chronic asymptomatic viral hepatitis is allowed.
* Positive test results from chronic hepatitis B infection (defined as positive HBsAg serology) and/or positive test results for hepatitis C (HCV antibody serology test).
* Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer currently in complete remission, or any other cancer from which the patient has been disease-free for 1 year
* Active central nervous system (CNS) malignancy or symptoms of CNS spread or administration of IT chemotherapy within 14 days prior to Day 1.
* Extramedullary disease causing symptoms and/or involving the CNS or spinal canal - asymptomatic extramedullary disease outside the CNS and spinal canal is eligible provided the marrow has measurable disease.
* Known autoimmune disease requiring active treatment with steroids or other immunosuppressive medications within 14 days before Cycle 1 Day. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Persons with a condition requiring systemic treatment with steroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before Cycle 1 Day 1.
* The potential risk of QT/QTc prolongation is unknown in humans receiving

TriKE therefore either of the following is an exclusion criteria:

* QTc interval > 480 msec at screening
* A family history of long QT syndrome
* Psychiatric illness/social situations that, in the judgement of the enrolling Investigator, would limit compliance with study requirements.
* Other illness or a medical issue that, in the judgement of the enrolling Investigator, would exclude the patient from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
MTD (ug/kg/day) | 6 months
  Maximum tolerated dose (MTD) of GTB-3650 TriKE defined as the dose level that most closely corresponds to the target dose limiting toxicity (DLT) proportion of 20% or less.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Feasibility ofGTB-3650 TriKE. | 6 months
  Evaluate the safety and feasibility of GTB-3650 TriKE repeat dosing based on the incidence of adverse events (AEs) using CTCAE v5 grading unless otherwise indicated.
Event free survival | 6 months
  Event free survival (EFS) defined as time to death, relapse after a complete remission (CR), or progression (no remission and requires a change in therapy for disease control)
Overall survival (OS) | 6 months
  Overall survival (OS) at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States